CLINICAL TRIAL: NCT05016323
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel Groups, Phase II Clinical Trial to Evaluate the Efficacy and Safety of HR19042 Capsules in the Treatment of Primary IgA Nephropathy.
Brief Title: A Study to Evaluate the Efficacy and Safety of HR19042 Capsules in the Treatment of Primary IgA Nephropathy.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR19042-201
Record Dates: First submitted 2021-08-17; First posted 2021-08-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, multicenter, placebo-controlled, parallel groups, Phase II clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR19042 Capsules (Experimental)
  Interventions: Drug: HR19042 Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HR19042 Capsules — HR19042 Capsules
  Arms: HR19042 Capsules
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of HR19042 capsules compared to matching placebo for the treatment of primary IgA nephropathy, and explore the optimal dose for the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients ≥18 years old；
2. Biopsy-confirmed primary IgA nephropathy；
3. Urine protein≥0.75 g/24hr or urine protein creatinine ratio (UPCR)≥0.5 g/g；
4. Estimated GFR (using the CKD-EPI2009 formula) ≥30mL/min/1.73 m2；
5. Willing and able to take adequate contraception during the trial;
6. Willing and able to give informed consent and follow the protocols during the trial.

Exclusion Criteria:

1. Systemic diseases which could lead to secondary IgA nephropathy；
2. Patients with severe chronic infection or active infection under systemic antibiotic therapy in previous 14 days；
3. Patients with severe cardiovascular diseases；
4. Patients diagnosed with malignancy within the past 5 years；
5. Patients with liver cirrhosis；
6. Patients received organ transplantation；
7. Patients with uncontrolled Type 1 or 2 diabetes；
8. Positive results in HIV-Ab/TP-Ab/ HBsAg/HCV-Ab tests；
9. Patients treated with any systemic immunosuppressive drugs (excluding corticosteroids) within the past 12 months before screening；
10. Patients treated with any systemic corticosteroids within the past 3 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in urine protein creatinine ratio (UPCR) | 9 months

SECONDARY OUTCOMES:
Change from baseline in 24-hour proteinuria | 9 months
Change from baseline in urine albumin creatinine ratio (UACR) | 9 months
Change from baseline in estimated GFR | 9 months
Change from baseline in estimated GFR | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639